CLINICAL TRIAL: NCT01236131
Title: Characterization of Novel Organisms in the Genital Tract of Women With PID and Determination of Their Association With Endometritis.
Brief Title: The Role of Novel Organisms in Acute Endometritis
Status: Completed | Type: Observational
Sponsor: Sharon Hillier (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Hillier, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO10080491; 1U19AI084024-01 (NIH)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endometrial biopsy specimens and isolates may be retained and stored in various registries such as:
  1. Human Microbiome Project
  2. J Craig Venture Institute
  3. PathoGene
  4. American Type Culture Collection
  5. CGS MindTouch Wiki hosted on Amazon's Elastic Compute Cloud (http://www.amazon.com/gp/browse.html?node-3435361)52 and will utilize MindTouch's Amazon Machine Image of their Wiki platform for rapid deployment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endometrial biospy samples: The Endometrial Biopsy samples will be provided by women enrolled in the University of Pittsburgh IRB PRO10010112 and PRO10010159
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Not Applicable- no intervention

SUMMARY:
The goal of this project is to identify the microorganisms present in the endometrial samples obtained from women with or without evidence of endometritis using a combination of culture methods, rRNA sequencing and whole genomic sequencing. The overarching aim of these studies is to identify the etiology of endometritis. The investigators will define the role of fastidious anaerobic microorganisms in the etiology of PID, and assess whether antibiotic treatment regimens used for the treatment of PID have activity against the novel organisms linked with pelvic infections.

ELIGIBILITY:
Inclusion Criteria:

* This is a laboratory research study involving the use of biologic specimens only.
* Specimens (endometrial biopsy samples) collected from subjects who meet the inclusion criteria for PRO10010159 and PRO10010112 will be utilized for this study.

Exclusion Criteria:

* Specimens (endometrial biopsy samples) that are collected from subjects enrolled in PRO10010159 and PRO10010112 that are insufficient will not be included in this study.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Endometrial biopsy samples from women participating in University of Pittsburgh IRB PRO10010112 and PRO10010159
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2010-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Identification of Novel Organsims from PRO10010159 | 12 months after participant enrollment in PRO10010159
  This study will use optimized culture methods which can support the growth of fastidious organisms to describe the microorganisms in endometrial tissue samples obtained from the 200 women enrolled in the cervicitis cohort (PRO10010159, T Cell Response).
Identification of Novel Organisms from PRO10010112 | 30 days after participant enrollment in PRO10010112
  This study will use optimized culture methods which can support the growth of fastidious organisms to describe the microorganisms in endometrial tissue samples obtained from 250 women enrolled in the acute PID study before and after treatment (PRO10010112, Acute PID treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Research Institute, Pittsburgh, Pennsylvania, United States